CLINICAL TRIAL: NCT04811963
Title: SpO2 Accuracy Validation of the OxySoftN Sensor Via Reference CO-Oximetry in Healthy, Well-Perfused Subjects
Brief Title: SpO2 Accuracy Low Saturation Validation of the OxySoftN Sensor
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: MDT20028OXYLOV
Record Dates: First submitted 2021-03-12; First posted 2021-03-23 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Hypoxia; Desaturation of Blood
Keywords: Oxygen Saturation; Invasive Controlled Desaturation
MeSH Terms: conditions — Hypoxia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

INTERVENTIONS:
Device: Non-Invasive Controlled Hypoxia — Following arterial cannulation, hypoxia is induced by reducing the percent of inspired oxygen the subject breathes while simultaneous measurements are recorded from the test pulse oximeters and arterial blood samples are collected at targeted levels of saturation.
  Other Names: Desaturation; Blood Sampling

SUMMARY:
To compare prototype pulse oximeter saturation measurements, during normal to low saturation, to saturation measurements made by a multi-wavelength CO-oximeter, taken from arterial blood samples from healthy human subjects.

DETAILED DESCRIPTION:
The study utilizes a single-site, physiology laboratory (Clinimark) for non-randomized, prospective, observational studies. The goal is to enroll a minimum of ten subjects. Subjects may be of any race, ranging in pigmentation from light to dark to meet the study design requirements.

The general purpose of Invasive Controlled Desaturation Studies is to validate the SpO2 and pulse rate accuracy in comparison to reference-standard measurements of blood SaO2 by a CO-oximeter during low saturation conditions. This is achieved through paired observations of SpO2 and SaO2 values over the specified SpO2 accuracy range of 60 % to 100 % SaO22 of the prototype pulse oximeter on a group of healthy adult volunteers. The fraction of inspired oxygen (FiO2) delivered to test subjects is varied to achieve a series of targeted steady-state saturation periods. Arterial blood samples are periodically taken from an indwelling arterial catheter for use in the comparison.

Pulse rate accuracy will be evaluated during the same data collection period as SpO2. Pulse rate will be compared to reference ECG heart rate. In the unlikely event that the ECG monitor malfunctions, the Pulse rate reference may be taken using the average pulse rate value from the transfer standard pulse oximeters. This study is designed to support an FDA submission for pulse rate and saturation accuracy in a diverse subject population during low saturation conditions over a specified saturation range for the OxySoftN pulse oximetry system.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have the ability to understand and provide written informed consent
2. Adult subjects 18 to 50 years of age.
3. Subject must be willing and able to comply with study procedures and duration.
4. Subject is a non-smoker or who has not smoked within 2 days prior to the study.
5. Male or female of any race.
6. Cleared same day Health Assessment form and health screening.
7. Cleared physical exam by a licensed physician, physician assistant, or advanced practice nurse (medical exam includes 12-lead ECG, medical history and blood test to show no sickle cell disease present)
8. Successful Perfusion Index Ulnar/Ulnar+Radial Ratio test showing adequate collateral blood flow.

Exclusion Criteria

1. Subject is considered as being morbidly obese (defined as BMI >39.5)
2. Compromised circulation, injury, or physical malformation of fingers, hands, ears or forehead/skull or other sensor sites which would limit the ability to test sites needed for the study. (Note: Certain malformations may still allow subjects to participate if the condition is noted and would not affect the sites utilized.)
3. Females of childbearing potential, who are pregnant, who are trying to get pregnant or who have a urine test positive for pregnancy on the day of the study
4. Subjects with COHb levels >3% as assessed by CO-Oximetry during the procedure
5. tHb < 10 g/dl as assessed by CO-Oximetry during the procedure
6. MetHb ≥ 2% as assessed by CO-Oximetry during the procedure
7. Subjects with known respiratory conditions such as:

   1. uncontrolled / severe asthma,
   2. flu or influenza type infection
   3. pneumonia / bronchitis,
   4. shortness of breath / respiratory distress,
   5. unresolved respiratory or lung surgery,
   6. emphysema, COPD, lung disease
8. Subjects with known heart or cardiovascular conditions such as:

   1. Hypertension: systolic >140mmHg, or Diastolic >90mmHg on 3 consecutive readings.
   2. have had cardiovascular surgery
   3. Chest pain (angina)
   4. heart rhythms other than a normal sinus rhythm or
   5. with respiratory sinus arrhythmia
   6. previous heart attack
   7. blocked artery
   8. unexplained shortness of breath
   9. congestive heart failure (CHF)
   10. history of stroke
   11. transient ischemic attack
   12. carotid artery disease
   13. myocardial ischemia
   14. myocardial infarction
   15. cardiomyopathy
9. Self-reported health conditions as identified in the Health Assessment Form

   1. diabetes,
   2. uncontrolled thyroid disease,
   3. kidney disease / chronic renal impairment,
   4. history of seizures (except childhood febrile seizures),
   5. epilepsy,
   6. history of unexplained syncope,
   7. recent history of frequent migraine headaches,
   8. recent symptomatic head injury, within the last 2 months
   9. Subjects with known clotting disorders
   10. history of bleeding disorders or personal history of prolonged bleeding from injury
   11. history of blood clots
   12. hemophilia
   13. current use of blood thinner: prescription or daily use of aspirin
   14. Subjects with Severe contact allergies to standard adhesives, latex or other materials found in pulse oximetry sensors, ECG electrodes, respiration monitor electrodes or other medical sensors
   15. Subjects with prior or known severe allergies to lidocaine (or similar pharmacological agents, e.g. Novocain) or heparin
   16. Arterial cannulation within the last 30 days prior to study date, (this may exclude only one radial artery site. Left or right)
   17. History of clinically significant complications from previous arterial cannulation.
   18. A radial artery with ten or more arterial cannulations right or left, excludes that site.
   19. Unwillingness or inability to remove colored nail polish or colored artificial nails other than clear from test digits.
   20. Other known health condition, should be considered upon disclosure in Health Assessment form

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population includes a minimum of ten healthy non-smoking (or has refrained from smoking for 2 days) competent adults 18-50 years of age. The subject selection will be an equitable distribution of males and females of any race with at least 2 darkly pigmented subjects or 15% of the subject pool, whichever is larger.
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-04-09 (Actual)

PRIMARY OUTCOMES:
To investigate performance of the OxySoft device by measuring oxygen saturation accuracy over a Low Saturation range of 60-80% | April 2021
  To validate the proposed claims for saturation accuracy in a diverse subject population during Low Saturation over a specified saturation range. The acceptance criteria for the OxySoftN Sensor SpO2 during Low Saturation conditions across the saturation range of 60-80% when paired with the N-600x, PM1000N and Oxicable:
  SpO2 OxySoftN ± 3% (Arms)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Cabrera, MD, Principal Investigator — Clinimark, LLC
Locations (1):
- Clinimark, Louisville, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
All participant data will be analyzed and outlined in final study report. Individual participant data will only be made available to the participant and or participant primary care physician as applicable.